CLINICAL TRIAL: NCT02335996
Title: Impact Hypercortisolism on Adipose Epicardial and on Myocardial Function
Brief Title: Hypercortisolism and Epicardial Adipose Tissue
Acronym: Hyper-Cor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-23; 2014-A01302-45 (Registry Identifier: ANSM); RCAPHM14_0343 (Other: APHM)
Record Dates: First submitted 2015-01-02; First posted 2015-01-12 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Hypercortisolism
MeSH Terms: conditions — Cushing Syndrome | interventions — Blood Specimen Collection; Leptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients with active hypercortisolism (Active Comparator)
  Interventions: Biological: Blood samples for measuring adiponectin, leptin and omentin plasma; Device: MRI at 3 Tesla
- Patients in remission of their hypercortisolism after surgery (Active Comparator)
  Interventions: Biological: Blood samples for measuring adiponectin, leptin and omentin plasma; Device: MRI at 3 Tesla

INTERVENTIONS:
Biological: Blood samples for measuring adiponectin, leptin and omentin plasma
Device: MRI at 3 Tesla — Evaluation by MRI at 3 Tesla of the amount of ectopic fat heart, liver and pancréas and bone marrow.

SUMMARY:
Identifying hypercortisolism patients at risk for cardio-vascular events despite biological cure, and determine which patients should be particularly followed. Hypercortisolic patients represent an ideal in vivo model to determine the interactions between glucocorticoids and ectopic fat development.

ELIGIBILITY:
Inclusion Criteria:

* Major, male or female
* Introducing an active or healed hypercortisolism caused by Cushing's disease
* signed informed consent.

Exclusion Criteria:

* Elderly patients under 18 years
* Pregnant or lactating women
* Previous history of myocardial infarction
* Antecedent congenital cardiomyopathy
* Adrenocorticotropic hormone-independent Hyperadrenocorticism
* Hyperadrenocorticism by ectopic Adrenocorticotropic hormone secretion
* Treatment with corticosteroids or insulin
* Specific contraindication to the achievement of Nuclear Magnetic Resonance (metal heart valves, pacemakers, metallic foreign body, claustrophobia)
* Persons deprived of liberty
* Persons not affiliated to a social security scheme
* People unable to give their consent in writing (in person or with the assistance of a third party).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
measuring the volume of epicardial adipose tissue, as measured by MRI to 3 Tesla. | 36 months
Assess insulin resistance by the blood sugar and insulin levels | 36 months
Assess cardiovascular risk by a blood complete lipid profile | 36 months

SECONDARY OUTCOMES:
Assess insulin resistance by the blood leptin, adiponectin and omentin plasma level | 36 months
Assess cardiovascular risk by the blood leptin, adiponectin and omentin plasma level | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Director, Study Director — Asistance Publique Hôpitaux Marseille
Locations (1):
- Assistance Publique Hôpitaux Marseille, Marseille, France